CLINICAL TRIAL: NCT05377034
Title: A Multinational, Double-blind, Placebo-Controlled, Parallel Randomized Arms, Phase II Trial to Compare Safety and Efficacy of Selective Internal Radiation Therapy (Y-90 Resin Microspheres) Followed by Atezolizumab Plus Bevacizumab) Versus Selective Internal Radiation Therapy (SIRT-Y90) Followed by Placebo in Patients With Locally Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Multinational Phase II Trial to Compare Safety and Efficacy of SIRT (Y-90 Resin Microspheres) Followed by Atezolizumab Plus Bevacizumab, vs SIRT (SIRT-Y90) Followed by Placebo in Locally Advanced HCC Patients
Acronym: STRATUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Hoffmann-La Roche (Industry); Sirtex Medical (Industry); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHCC09 STRATUM
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Hepatocellular Carcinoma
Keywords: SIRT-Y90; Atezolizumab plus Bevacizumab; Hepatocellular Carcinoma; SIR-Sphere
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed in a double-blind manner. The investigators, monitoring team, site staff, and all patients will be blinded to the study treatments from the time of randomization until database lock. Biostatisticians involved in preparing the randomization and safety data analysis for Data and Safety Monitoring Board (independent to study statistician) will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): SIRT-Y90 + 1200mg atezolizumab + 15mg/kg bevacizumab
  Interventions: Combination Product: SIRT-Y90 with Atezolizumab + Bevacizumab
- Control Arm (Experimental): SIRT-Y90 + placebos (IV)
  Interventions: Combination Product: SIRT-Y90 with Placebo (IV)

INTERVENTIONS:
Combination Product: SIRT-Y90 with Atezolizumab + Bevacizumab — Single or two-staged delivery of SIRT-Y90 (4 to 6 weeks), followed by 1200mg atezolizumab + 15mg/kg bevacizumab administered by IV at every 3 weeks for 18 months.
  Arms: Study Arm
Combination Product: SIRT-Y90 with Placebo (IV) — Single or two-staged delivery of SIRT-Y90 (4 to 6 weeks), followed by placebo at every 3 weeks for 18 months.
  Arms: Control Arm

SUMMARY:
This is a multi-national, phase II, parallel-arm, double-blind, placebo-controlled, two-arm study designed to assess the efficacy and safety of SIRT-Y90 followed by atezolizumab plus bevacizumab [study arm], versus SIRT-Y90 followed by placebo [control arm] in patients with locally advanced Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
This study will enroll 100 patients randomized in a 1:1 allocation ratio (50 in each arm) to one of the two arms.

* Study arm: SIRT-Y90 + 1200mg atezolizumab + 15mg/kg bevacizumab
* Control arm: SIRT-Y90 + placebos (IV)

The patients will be recruited from up to 15 sites from the Asia-Pacific Hepatocellular Carcinoma (AHCC) Trials Group (subjected to feasibility studies and ethics approval). Proposed sites are in Singapore, China, South Korea, and Taiwan.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for this study:

1. Unequivocal diagnosis of HCC (AASLD 2010 diagnostic criteria or histology) that is locally advanced without extra-hepatic metastases but with significant tumor burden, i.e.,

   * Tumor confined to the liver that is beyond the up-to-7 criteria, and/or
   * Tumor with vascular invasion VP 1-3 and/or Vv 1-2 (at the discretion of site investigator) Both local and central assessments are required at screening, prior to any study treatment. Sites are required to send all CT/MRI images for central imaging review. The central assessment result will be made known to sites and will take precedence in determining a patient's study eligibility in case of a discrepancy between local and central review.
2. Aged 21 years old and above of either gender.
3. Patient eligible for SIRT-Y90 treatment after assessment with macro-aggregated albumin labeled with technetium-99 (Tc-99m MAA) scan on SPECT/CT or planar imaging with all of the following criteria prior to each SIRT-Y90 treatment:

   * Lung shunting <20% on SPECT/CT or planar imaging
   * Lung dose limit of <25Gy for single treatment or <30Gy for cumulative treatment (second delivery within 4-6 weeks)
4. No prior radiation to the liver.
5. No prior systemic adjuvant or neoadjuvant therapy for HCC.
6. Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with spiral CT scan or MRI.
7. Negative HIV test at screening, with the following exception - patients with a positive HIV test at screening are eligible provided they fulfil all of the following criteria:

   * Are stable on anti-retroviral therapy
   * Have a CD4 count ≥ 200/μL
   * Have an undetectable viral load
8. Documented virology status of hepatitis, as confirmed by screening hepatitis B virus (HBV) and hepatitis C virus (HCV) tests.
9. Patients with active HBV: HBV DNA <3000 IU/mL, initiation of anti-HBV treatment at least 14 days prior to randomization, and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir).

   For patients with HBV DNA ≥ 500 IU/mL during screening, anti-HBV treatment will be initiated and HBV DNA levels will be re-assessed prior to randomization.
10. ECOG performance status 0 - 1.
11. Child-Pugh A (up to 6 points).
12. Adequate hematological, renal, and hepatic function as follows:

    * Lymphocyte count ≥ 0.5 x 10**9/L (500/μL)
    * Platelets ≥75,000/μL without transfusion
    * Hemoglobin >9.5 g/dL (Patients may be transfused to meet this criterion.)
    * Serum bilirubin ≤ 3 x ULN
    * For patients not receiving therapeutic anticoagulation: INR and aPTT ≤ 2.0 x ULN
    * ALP ≤5×institutional upper limit of normal
    * AST and ALT ≤5×institutional upper limit of normal
    * Albumin ≥2.8 g/dL
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 30 mL/min (calculated using the Cockcroft-Gault formula)
    * Absolute Neutrophil Count ≥1.5×10**9/L without granulocyte colony-stimulating factor support
    * Urine dipstick for proteinuria <2+ at screening

      * Patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1g of protein in 24 hours
13. Life expectancy of at least 3 months without any active treatment.
14. Suitable for protocol treatment as determined by clinical assessment undertaken by the site investigator.
15. Performance of an esophagogastroduodenoscopy (EGD) within 6 months prior to randomization as part of pre-procedure work-up or during screening, and assessment and complete treatment of varices of all sizes per local standard of care prior to randomization.

    Patients with varices should be re-assessed prior to randomization to ensure complete treatment of varices of all sizes per local standard of care.
16. Willing, able and mentally competent to provide written informed consent prior to any testing undertaken for this study protocol, including screening tests and evaluations that are not considered to be part of the patient's routine care.
17. Female patients must be either postmenopausal or, if premenopausal, must have a negative pregnancy test and agree to use two forms of contraception if sexually active during the treatment period, for at least 5 months after the last dose of atezolizumab and 6 months after the last dose of bevacizumab.
18. Male patients must be surgically sterile, or if sexually active and having a pre-menopausal female partner, they must be using an acceptable form of contraception during the treatment period and for 6 months after the last dose of bevacizumab.

Exclusion Criteria:

The following criteria should be checked. If ANY apply, the patient must not be included in the study:

1. Patient not eligible for SIRT-Y90 treatment after assessment with macro-aggregated albumin labeled with technetium-99 (MAA) scan on SPECT/CT or planar imaging.
2. Patients who have SAE > grade 3 within 4 weeks after receiving SIRT-Y90. For patients who experience SAE > grade 3 after receiving SIRT-Y90 (1st or 2nd administration), the duration between the SIRT-Y90 dose and randomization and/or 1st and 2nd SIRT-Y90 dose (for two-staged delivery) may be extended by an additional 4 weeks to re-assess the patient's eligibility.
3. Patients who have had >2 administrations of hepatic artery directed therapy.
4. Patients who have had hepatic artery directed therapy done <4 weeks prior to date of ICF signing.
5. Patients who have had systemic adjuvant or neoadjuvant therapy for HCC.
6. Prior hepatic radiation therapy for HCC or other malignancy.
7. Patient who has received any immunotherapy (including interferon-alfa, peginterferon alfa-2a, peginterferon alfa-2b, thymosin-α1, etc.) within 30 days prior to randomization, is currently receiving immunotherapy or is planned to start immunotherapy during the study (e.g., for the management of active CHB or CHC according to local guidelines).
8. Has evidence that <30% of the total liver volume is disease-free.
9. Currently receiving any other investigational agents for the treatment of their cancer.
10. Has intractable clinical ascites (in spite of optimal diuretic treatment) or any other clinical signs of liver failure, on physical examination.
11. Untreated or incompletely treated esophageal and/or gastric varices prior to randomization.
12. Presence of tumor thrombus in the main trunk of the portal vein or a portal vein branch contralateral to the primarily involved lobe (or both) i.e. beyond VP3 and/or tumor thrombus in the inferior vena cava or right atrium i.e. beyond Vv2.
13. Any metastatic disease i.e. lymph node ≥15 mm in short axis or distant metastasis.
14. Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
15. Presence of clinical signs of CNS metastases due to their poor prognosis and because progressive neurologic dysfunction would confound the evaluation of neurologic and other adverse events.
16. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection (except viral hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
17. Inadequately controlled arterial hypertension (defined as systolic blood pressure [BP]>150 mmHg and/or diastolic BP >100 mmHg), based on an average of at least three BP readings on separate occasions.

    • Anti-hypertensive therapy to achieve these parameters is allowed.
18. Any of the following contraindications to angiography and selective visceral catheterization:

    * Bleeding diathesis, not correctable by the standard forms of therapy.
    * Severe peripheral vascular disease that would preclude arterial catheterization.
19. Significant cardiovascular disease (such as cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to randomization), unstable arrhythmia, or unstable angina.
20. History of congenital long QT syndrome or corrected QT interval > 500 ms (calculated with use of the Fridericia method) at screening
21. History of uncorrectable electrolyte disorder affecting serum levels of potassium, calcium, or magnesium
22. Current or recent use (within 10 days prior to angiogram) of aspirin (>325 mg/day) or current or recent treatment with dipyridamole, ticlopidine, clopidogrel, and cilostazol.

    • Use of dipyridamole, ticlopidine, clopidogrel, and cilostazol is allowed for patients who do not have any active bleeding for the past 6 months after review with attending physician.
23. Current or recent (within 10 days prior to angiogram) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose.

    * Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR <1.5×ULN and aPTT is within normal limits (according to institutional standards) within 14 days prior to Day 1 of Cycle 1.
    * Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
24. History of allergic reactions attributed to compounds of similar chemical or biologic composition to SIRT-Y90 or atezolizumab or bevacizumab.
25. The patient has active or history of autoimmune disease or immune deficiency such as, but not limited to, multiple sclerosis, systemic lupus erythematosus, and inflammatory bowel disease, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months prior to screening.
26. The patient requires concomitant treatment with any immunosuppressive or immunostimulant agent, or with systemic corticosteroids prescribed for chronic treatment (more than 7 consecutive days).
27. Inability or unwillingness to understand or sign a written informed consent document.
28. Female patients who are pregnant or currently breastfeeding.
29. Current enrolment in any other investigational therapeutic drug or device study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (BORR) at 9 months post-randomization. | 9 months post-randomization.
  The number of patients whose Best Overall Response (BOR) at 9 months post-randomization is a partial response or complete response per RECIST v1.1 and mRECIST, divided by the total number of patients in the analysis population.

SECONDARY OUTCOMES:
Best Overall Response Rate (BORR) at 12-months and 18-months post-randomization. | 12 months and 18 months post-randomization.
  The number of patients whose Best Overall Response (BOR) at 12 and 18 months post-randomization is a partial response or complete response per RECIST v1.1 and mRECIST, divided by the total number of patients in the analysis population.
Sustained response rates at 9, 12 and 18 months. | 9,12 and 18 months post-randomization.
  The number of patients whose BOR at time t (t = 9, 12 and 18 months) is a partial response or complete response confirmed on a subsequent visit by CT scan, divided by the total number of patients in the analysis population.
Disease control rates at 9, 12 and 18 months. | 9,12 and 18 months post-randomization.
  The number of patients whose BOR at time t (t = 9, 12 and 18 months) is a partial response, complete response, or stable disease per RECIST v1.1 and mRECIST, divided by the total number of patients in the analysis population.
Time to response. | Up to 19 months post-randomization.
  The time between randomization and the date of first partial response or complete response. For those who have no partial response or complete response by the time of analysis will be censored on the date of last evaluable tumor assessment on or before the time of analysis or the end of study treatment, whichever is earlier.
Duration of response (DOR). | Up to 19 months post-randomization.
  DOR is the time from the date of first partial response or complete response to date of tumor progression or death from any cause, whichever is earlier. For those who are alive and have not experienced disease progression by the time of analysis will be censored on the date of last evaluable tumor assessment on or before the time of analysis or the end of study treatment, whichever is earlier.
Time to disease progression. | Up to 19 months post-randomization.
  The time between randomization and the date of tumor progression at any site in the body or death due to HCC. For those who remain alive or died due to other reasons or have not experienced disease progression, time to disease progression will be censored on the date of last evaluable tumor assessment on or before the time of analysis or the end of study treatment, whichever is earlier.
Progression-free survival (PFS). | Up to 19 months post-randomization.
  The time from randomization to the date of tumor progression at any site in the body or death from any cause, whichever is earlier. For those who remain alive and have not progressed, PFS will be censored on the date of the last evaluable tumor assessment on or before the time of analysis or the end of study treatment, whichever is earlier. Progression-free survival rates will also be calculated at time t (t = 12 and 18 months).
Overall survival (OS). | 12 and 18 months post-randomization.
  The time from randomization to death from any cause. Patients who are alive will be censored at the last date the patient was known to be alive on or before the time of analysis. Overall survival rates will also be calculated at time t (t = 12 and 18 months).
EQ-5D-5L utility index at 12 and 18 months. | 12 and 18 months post-randomization.
  The EQ-5D-5L utility index will be calculated using the EQ-5D-5L value set for the recruiting site country (Singapore, China, South Korea, and Taiwan) based on EQ-5D-5L assessment at time t (t = 12 and 18 months). Currently, there is no value set available for Singapore. However, if it will not be available by the time of the analysis, another suitable country's value set will be used. The EQ-VAS will also be used as an additional measure.
FACT-Hep scores at 12 and 18 months. | 12 and 18 months post-randomization.
  The FACT-Hep total score along with subscales (physical well-being, social/family well-being, emotional well-being, functional well-being, hepatobiliary cancer, trial outcome index, FACT-G total score) will be calculated using the FACT-Hep (version 4) scoring guideline based on FACT-Fep assessment at time t (t = 12 and 18 months).
Quality-adjusted life years at 18 months. | 18 months post-randomization.
  The quality-adjusted life-years (QALYs) will be calculated as the area under the EQ-5D-5L index during the 18 months.

OTHER OUTCOMES:
SIRT-Y90 post-treatment dosimetry. | 4-week SIRT pre-randomization; 3, 6, 12 and 18 months post-randomization.
  Voxel-level mean tumor absorbed dose (Dmean) and mean biological effective dose (BEDmean) for SIRT-Y90 will be calculated using CT images using local deposition method. In addition, administered activity and mean absorbed dose to treated liver volume (including both tumoral and non-tumoral tissue) will be used as dosimetry parameters. Dose response evaluation will be attempted based on the information obtained and follow-up anatomical evaluation. The impact of tumour absorbed dose on BORR, tumour response as assessed by RECIST v1.1 and mRECIST and outcomes of patients receiving SIRT-Y90 (3, 6, 12 and 18 months) will be assessed.
Hepatic progression-free survival (HPFS). | Up to 19 months post-randomization.
  Hepatic progression-free survival (HPFS) is defined as the time from randomization and the date of tumor progression in liver or death from any cause, whichever is earlier. For those who remain alive and have not progressed in the liver, HPFS will be censored on the date of the last evaluable tumor assessment on or before the time of analysis or end of study treatment, whichever is earlier.
Tumor resectability rates at 12 and 18 months. | 12 and 18 months post-randomization.
  Tumor resectability rate at time t (t = 12 and 18 months) is defined as the number of patients undergone surgical resection for the target lesions of HCC by time t, divided by the total number of patients in the analysis population.
Impact of Albumin-Bilirubin (ALBI) grade on the overall survival and progression-free survival outcomes of HCC patients undergoing SIRT-Y90. | Up to 19 months post-randomization.
  The ALBI (Albumin-Bilirubin) score is calculated based on serum albumin and bilirubin levels and values are classified into three ALBI grades: Grade 1, Grade 2 and Grade 3, where Grade 1 indicates a better outcome. In this trial, the ALBI grade at screening will be correlated to information obtained during treatment and follow up visits such as clinical outcomes like mortality, grade 3 or 4 adverse events and/or radiological responses as measured by RECIST v1.1 and mRECIST.
Occurrence of adverse events and adverse events related to study treatment. | Up to 19 months post-randomization.
  Occurrence of adverse events and adverse events related to study treatment up to 30 days post last study treatment dose, including abnormal hematological and biochemical parameters.
Occurrence of ≥3 grade adverse events (graded with NCI CTCAE v5.0). | Up to 19 months post-randomization.
  Occurrence of ≥3 grade adverse events (graded with NCI CTCAE v5.0) up to 30 days post last study treatment dose, including abnormal hematological and biochemical parameters.
Occurrence of adverse events of special interest. | Up to 21 months post-randomization.
  Occurrence of adverse events of special interest up to 90 days post last study treatment dose, including abnormal hematological and biochemical parameters.
Occurrence of adverse events leading to study treatment discontinuation or interruption. | Up to 18 months post-randomization.
  Occurrence of adverse events leading to study treatment discontinuation or interruption.
Occurrence of serious adverse events after initiation of study treatment until 90 days post last study treatment dose. | Up to 21 months post-randomization.
  Occurrence of serious adverse events after initiation of study treatment until 90 days post last study treatment dose.
Occurrence of adverse events leading to death. | Up to 21 months post-randomization.
  Occurrence of adverse events leading to death.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce CHOW, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (14):
- China (4):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - People's Liberation Army General Hospital (1st and 6th Medical Centre), Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Shandong Cancer Hospital, Jinan
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided